CLINICAL TRIAL: NCT05900843
Title: Prevalence and Correlations of Weight Abnormalities With Diet and Exercise Frequency in Egyptian Children With Cerebral Palsy
Brief Title: Weight Abnormalities With Diet and Exercise Frequency in Egyptian Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tayseer Saber Abdeldayem, Lecturer, Beni-Suef University
Other Study IDs: P.T.REC/012/004234
Record Dates: First submitted 2023-02-03; First posted 2023-06-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Obesity, Childhood; Cerebral Palsy; Weight, Body; Abdominal Obesity
Keywords: weight abnormalities; abdominal obesity; cerebral palsy
MeSH Terms: conditions — Pediatric Obesity; Cerebral Palsy; Body Weight; Obesity, Abdominal

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study was to find prevalence and correlations of different weight abnormalities and risk of abdominal obesity in a random sample of Egyptian children suffering from cerebral palsy. This cross- sectional study hypothesize the prevalence of weight abnormalities and risk of abdominal obesity in addition to positive correlations between weight abnormalities and number of exercise hours and frequency of meals in a random sample of Egyptian children suffering from cerebral palsy

RESEARCH QUESTION:

1. What is the prevalence of weight abnormalities and and risk of abdominal obesity in Egyptian children with cerebral palsy?
2. Does the weight abnormalities correlates with number of exercise hours or frequency of meals in children with cerebral palsy?

DETAILED DESCRIPTION:
This cross- sectional study will be conducted to identify the prevalence of weight abnormalities and risk of abdominal obesity in a random sample of Egyptian children suffering from cerebral palsy. It included all cerebral palsy cases at six private pediatric rehabilitation clinics in four different governorates (Cairo, Alexandria, Sharkia and Beni-Suef). Data will be collected from patients, records of the referrals to pediatric physical therapy rehabilitation clinics and measurements of weight, height, waist circumference and hip circumference performed by the therapist.

These six settings were selected because;1) They represent different geographical and socioeconomic levels in Egypt, 2) All of them offer pediatric physical therapy rehabilitation sessions at approximately the same range of price ,3) At that time general hospitals were still strictly committed to corona virus control measures, so no data could be available from general hospitals.

The following information will be extracted from the patient records: Sex, Age, Diagnosis, subtype of Cerebral Palsy, level of function and degree of spasticity., associated impairments, dietary intake (number of meals or quality of meals) and number of exercise hours per week. A questionnaire will be designed to get the care givers' report about presence of associated impairments, number of meals per day and number of exercising hours per week, type of associated impairments, quality of meals and type of exercises. All care givers of children diagnosed by cerebral palsy will be interviewed by the therapist to help them fill in the questionnaire and to obtain a consent of their participation. BMI; kg/m2 will be calculated by measuring height and weight. WHR will be calculated by measuring waist circumference and hip circumference. BMI and WHR percentiles will be reported according to sex-specific age group standards for growth set by the WHO growth charts.

ELIGIBILITY:
Inclusion Criteria:

* all children diagnosed as Cerebral Palsy between the age of 2 to 18 years old from both sexes in the participating clinics

Exclusion Criteria:

* Children suffering from developmental motor delays due to any other diagnosis
* Children who refused to engage in measurement procedures (weight, height, waist circumference and hip circumference)
* Children suffered from fixed deformity that didn't allow to get accurate measurements

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed as Cerebral Palsy between the age of 2 to 18 years
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 2 months
  weight and height are measured and compared to charts

SECONDARY OUTCOMES:
Exercising habits | 2 months
  number of exercise hours per week
Dietary habits | 2 months
  Number of meals per day

CONTACTS AND LOCATIONS:
Overall Officials: Sabah M Elkady, PhD, Study Chair — Cairo University; Mai A Ahmed, PhD, Study Chair — Beni-Suef University
Locations (1):
- Tayseer Saber Abdeldayem, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided